CLINICAL TRIAL: NCT04547088
Title: Efficacy and Safety of Camrelizumab Combined With Apatinib in Patients With First-line Platinum-resistant Recurrent/Metastatic Nasopharyngeal Carcinoma: a Single-center, Single-arm, Phase 2 Trail
Brief Title: Camrelizumab Combined With Apatinib in Patients With First-line Platinum-resistant Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-FXY-176
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Apatinib (Experimental): Patients with recurrent or metastatic nasopharyngeal carcinoma who failed to first-line platinum-based chemotherapy. Every patient will receive Apatinib 250mg orally every day and Camrelizumab 200mg iv every 3 weeks until disease progression or intolerance of side effects.
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — Anti-PD-1 targeted immunotherapy
  Other Names: SHR-1210
Drug: Apatinib — A small-molecule vascular endothelial growth factors receptor (VEGFR) tyrosine kinase inhibitor
  Other Names: Apatinib Mesylate

SUMMARY:
The purpose of this study is to explore the efficacy and safety of a combination of Camrelizumab and Apatinib regimen in treating recurrent or metastatic nasopharyngeal carcinoma patients who have failed first-line platinum-based chemotherapy.

DETAILED DESCRIPTION:
Currently, there is still no uniform treatment regimen in treating recurrent or metastatic nasopharyngeal carcinoma patients who failed to first-line platinum-based chemotherapy. Anti-PD-1 monoclonal antibody showed efficacy and safety in previous studies, however, the efficacy of immunotherapy alone was limited. Immunotherapy combined with other treatment regimens for recurrent or metastatic nasopharyngeal carcinoma is a strategy that needs to be urgently explored. Vascular endothelial growth factor (VEGF) is an important target in the treatment of nasopharyngeal carcinoma. Apatinib, a small-molecule tyrosine kinase inhibitor selectively inhibits vascular endothelial growth factor receptor 2 (VEGFR-2), has shown strong clinical utility. Previous clinical studies have confirmed that apatinib shows antitumor activity and tolerable toxicity in recurrent or metastatic nasopharyngeal carcinoma. Tumor vascular normalization and immune reprogramming interact synergistically and could enter a mutually reinforcing virtuous cycle by improving tumor microenvironment. The current national comprehensive cancer network (NCCN) guidelines also recommend Nivolumab and Pembrolizumab as a second-line treatment for recurrent or metastatic nasopharyngeal carcinoma. More and more evidence show that immunotherapy combined with anti-angiogenesis therapy has a synergistic effect, and Camrelizumab combined with apatinib therapy has achieved the initial effect in solid tumors. Based on this, this study aims to evaluate the efficacy and safety of Camrelizumab combined with apatinib in the patients with recurrent or metastatic nasopharyngeal carcinoma who failed to first-line platinum-based chemotherapy, to provide new evidence for individualized comprehensive treatment in nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed with recurrent or metastatic nasopharyngeal carcinoma which is not amenable to curative treatment with surgery and/or radiation therapy.
2. Age ≥ 18 years and ≤ 75 years, both genders.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
4. The life expectancy of at least 3 months.
5. Have failed for first-line platinum-based chemotherapy.
6. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
7. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment) as determined by:

   Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9 g/dL; serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), (for subjects with liver metastases, TBIL ≤3×ULN; ALT and AST≤5×ULN); Creatinine ≤1.5×ULN or creatinine clearance rate≥50 ml/min (Cockcroft-Gault formula); serum albumin ≥28 g/L; Thyroid-stimulating hormone (TSH) levels ≤1×ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤1× ULN may be enrolled); INR, APTT≤1.5 x ULN.
8. All women with fertility potential must undergo a urine or serum pregnancy test during screening and the results are negative.
9. Written informed consent.

Exclusion Criteria:

1. Known history of hypersensitivity to any components of the Camrelizumab formulation, or other monoclonal antibodies.
2. Prior exposure to immune checkpoint inhibitors, including anti-PD-1, anti-PD-L1, anti-PD-L2 antibodies.
3. Prior therapy with tyrosine kinase-inhibitor agent targeting at VEGFR.
4. There was a history of severe bleeding, and any bleeding events with a serious grade of 3 or more in CTCAE5.0 occurred within 4 weeks before screening.
5. Before treatment, MRI showed that the tumor may have invaded important blood vessels (such as enclosing the internal carotid artery/ vein), nasopharyngeal necrosis or researchers have determined that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during treatment.
6. Patients with abnormal blood coagulation and bleeding tendency (14 days before signing informed consent: INR is within the normal range without anticoagulant); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues. On the premise that the INR < 1.5, low-dose warfarin (1mg orally, once a day) or low-dose aspirin (daily dose not more than 100mg) is allowed for preventive purposes.
7. Arteriovenous thrombosis occurred within one year before the screening, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by intravenous catheterization due to early chemotherapy) and pulmonary embolism.
8. Patients with hypertension who cannot be well controlled by antihypertensive therapy (systolic blood pressure ≥ 140mmHg, diastolic blood pressure ≥ 90mmHg); patients with a history of hypertensive crisis or hypertensive encephalopathy.
9. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
10. Received any CYP3A4 inhibitor within 2 weeks before the first administration.
11. Have a history of Crohn's disease, ulcerative colitis, and chronic diarrhea.
12. Have a history of gastrointestinal perforation or fistula.
13. Any factors that affect oral drug.
14. Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
15. Join another clinical study at the same time, received any research drug within 4 weeks before the first administration of the drug.
16. Patients with any active autoimmune disease or a documented history of autoimmune disease such as pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
17. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
18. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease.
19. Be known to have active tuberculosis.
20. Hepatitis B virus (HBV) >2000 IU/ml or DNA ≥ 1×10^4/ml; or hepatitis C virus (HCV) RNA ≥ 1×10^3/ml).
21. Has an active infection requiring systemic therapy.
22. Has known active central nervous system metastases.
23. Severe, uncontrolled angiocardiopathy (heart failure > class II NYHA, unstable angina, myocardial infarction within past 1 year, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.).
24. Have been vaccinated with anti-tumor vaccines or have been vaccinated with live vaccines within 4 weeks before screening.
25. Pregnant or nursing.
26. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI)

SECONDARY OUTCOMES:
Disease control rate | 2 years
  A disease control rate is defined as either a confirmed CR or a PR or a SD, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI).
Duration of response | 2 years
  Defined from date of first confirmed CR or a PR to date of first documentation of progression or death due to any cause, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI).
Progression-free survival rate | 2 years
  Defined from date of registration to date of first documentation of progression or death due to any cause.
Overall survival rate | 2 years
  Defined from date of registration to date of first documentation of death from any cause or censored at the date of the last follow-up.
Incidence rate of adverse events (AEs) | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) as assessed by CTCAE v5.0.
PD-L1 expression on tumor and immune cells | 2 years
  The efficacy of the combination of Camrelizumab and apatinib as measured by objective response, will be described in patients according to PD-L1 positive and PD-L1 negative.
VEGFR-2 expression in tumor | 2 years
  The impact of VEGFR-2 on efficacy of the combination of Camrelizumab and apatinib will be explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Lan CY, Wang Y, Xiong Y, Li JD, Shen JX, Li YF, Zheng M, Zhang YN, Feng YL, Liu Q, Huang HQ, Huang X. Apatinib combined with oral etoposide in patients with platinum-resistant or platinum-refractory ovarian cancer (AEROC): a phase 2, single-arm, prospective study. Lancet Oncol. 2018 Sep;19(9):1239-1246. doi: 10.1016/S1470-2045(18)30349-8. Epub 2018 Aug 3. PMID 30082170
- [Background] Reck M, Mok TSK, Nishio M, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Lee A, Coleman S, Deng Y, Kowanetz M, Shankar G, Lin W, Socinski MA; IMpower150 Study Group. Atezolizumab plus bevacizumab and chemotherapy in non-small-cell lung cancer (IMpower150): key subgroup analyses of patients with EGFR mutations or baseline liver metastases in a randomised, open-label phase 3 trial. Lancet Respir Med. 2019 May;7(5):387-401. doi: 10.1016/S2213-2600(19)30084-0. Epub 2019 Mar 25. PMID 30922878
- [Background] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Derived] Yuan L, Jia GD, Lv XF, Xie SY, Guo SS, Lin DF, Liu LT, Luo DH, Li YF, Deng SW, Guo L, Zeng MS, Cai XY, Liu SL, Sun XS, Li XY, Li SC, Chen QY, Tang LQ, Mai HQ. Camrelizumab combined with apatinib in patients with first-line platinum-resistant or PD-1 inhibitor resistant recurrent/metastatic nasopharyngeal carcinoma: a single-arm, phase 2 trial. Nat Commun. 2023 Aug 14;14(1):4893. doi: 10.1038/s41467-023-40402-x. PMID 37580352